CLINICAL TRIAL: NCT05683444
Title: Octreotide Improves Human Lymphatic Fluid Transport a Translational Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Aarhus (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Thomas Holm-Weber, Medical Doctor, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P-2020-592
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Lymphatic Diseases; Chylothorax
MeSH Terms: conditions — Lymphatic Diseases; Chylothorax

STUDY DESIGN:
Intervention Model Description: Double-blinded cross over study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither the participant nor investigator nor outcomes assessor was aware of whether saline or octreotide was infused on the day of investigation and data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy participant 1 (Other)
  Interventions: Drug: Octreotide infusion; Drug: Saline infusion
- Healthy participant 2 (Other)
  Interventions: Drug: Octreotide infusion; Drug: Saline infusion

INTERVENTIONS:
Drug: Octreotide infusion — Octreotide infusion for 2,5 hours. 300 ng/kg/min bolus was given for the first 15 minutes and then a continuous infusion of 100 ng/kg/min for the remaining 135 minutes.
Drug: Saline infusion — Saline Infusion

SUMMARY:
This study aims to investigate whether octreotide, a medication used off-label to treat chylothorax, has a direct effect on human lymphatic drainage. To study the effects of octreotide, the researchers conducted a pre-clinical experiment using human lymphatic vessels mounted in a myograph chamber and a clinical experiment in which a double-blinded, randomized, cross-over trial was conducted in 16 healthy adults. The results of the study will be used to determine the role of octreotide in the treatment of chylothorax and other lymphatic disorders.

DETAILED DESCRIPTION:
This study aimed to investigate whether octreotide, a medication used off-label to treat chylothorax, has a direct effect on human lymphatic drainage. Chylothorax is a condition in which there is an accumulation of lymphatic fluid in the chest cavity, and the mechanism through which octreotide helps to resolve this condition is not well understood. It has been speculated that the drug may reduce lymph production, but this has not been directly demonstrated. To study the effects of octreotide on human lymphatic vessels, the investigators conducted two experiments: a pre-clinical experiment using human lymphatic vessels mounted in a myograph chamber, and a clinical experiment in which a double-blinded, randomized, cross-over trial was conducted in 16 healthy adults, assessed by using plethysmography and near-infrared fluorescence imaging. The results of the study will be used to determine the role of octreotide in the treatment of chylothorax and to clarify the mechanism through which it acts. It is important to continue researching and developing effective treatments for chylothorax, as it can be a difficult condition to manage and may cause serious complications if left untreated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* No daily medication (except birth control), or allergies towards contrast agents.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Lymph rate | During infusion
  Propulsions /minute
Lymph Pressure | During infusion
  mmHg assessed by near-infra fluorescence imaging
Capillary filtration rate | During infusion
  assessed by plethysmography
Capillary filtration coefficiency | During infusion
  assessed by plethysmography
Isovolumetric pressure | During infusion
  assessed by plethysmography

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: Undecided